CLINICAL TRIAL: NCT00008801
Title: hOKT3gamma1 (Ala-Ala) for the Prevention of Human Islet Allograft Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCRR-M01RR00400-0672
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-11-01 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Mellitus, Insulin-Dependent; Diabetes Mellitus, Experimental; Transplantation, Homologous; Islets of Langerhans Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Experimental | interventions — teplizumab

INTERVENTIONS:
Drug: hOKT3gamma1 (Ala-ala)

SUMMARY:
The broad, long-term goal of this proposal is to improve the results and applicability of islet allotransplantation early in the course of type 1 diabetes through the administration of selective and short-term immunotherapy. More specifically, the objectives of these studies is to conduct an open-labeled, one-year follow-up Phase I/II study in patients with surgical and type 1 diabetes to determine the safety, tolerability, immune activity, and pharmacokinetics of hOKT3gamma1 (Ala-ala) administration for the prevention of autoimmune destruction and rejection of allogeneic islet transplants.

DETAILED DESCRIPTION:
Adverse events will be monitored and recorded throughout the first year post-transplant. The proportion of surgical and type 1 diabetic subjects receiving an islet allotransplant who achieve and maintain full or partial islet graft function during the first year post-transplant will be determined to assess the efficacy of hOKT3gamma1 (Ala-ala) administration. Successful completion of the proposed clinical trial will increase our understanding of the safety, efficacy and underlying mechanisms of selective immunotherapy with the anti-CD3 monoclonal antibody hOKT3gamma1 (Ala-ala) for the maximization of engraftment and functional survival of allogeneic human islets in surgical and type 1 diabetic recipients.

ELIGIBILITY:
Inclusion:

* Primary islet allotransplant
* surgical or type 1 diabetes mellitus, complicated by signs and symptoms that persist despite intensive efforts made in close cooperation with their diabetes care team
* Age 18 or older
* must give written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States